# Statistical analysis plan (SAP)

# NCT03531463

Nordic Innovative Trials to Evaluate osteoPorotic Fractures (NITEP) Collaboration: The Nordic DeltaCon Trial protocol—non-operative treatment versus reversed total shoulder arthroplasty in patients 65 years of age and older with a displaced proximal humerus fracture: a prospective, randomised controlled trial

# **SECTION 1: ADMINISTRATIVE INFORMATION**

**Trial registration:** The trial is registered at <u>www.clincaltrials.gov</u> with the number NCT03531463.

**Protocol version:** This document has been written based on the information contained in the trial protocol published in BMJ Open (1).

# Statistical Analysis Plan (SAP) revision history:

| SAP version | Section changed | Description and reason for change | Date changed |
|---|---|---|---|
| 1.0 | Initial draft | | |
| 1.1 | Analyses | specified | 7.2.24 |
| 1.2 | References | added | 19.2.24 |
| 1.3 | Final agreement of SAP | | 16.11.25 |

# Roles and responsibilities:

| Role | Name |
|---------------------|--------------------------------|
| SAP author | Antti Launonen, Tore Fjalestad |
| Senior statistician | Are Hugo Pripp |
| Study trialist | Aleksi Reito |
| Chief investigator | Antti Launonen |

# **Signatures:**

| Role | Name | Date | Signature |
|---------------------|----------------|------|-----------|
| SAP author | Tore Fjalestad | | |
| Senior statistician | Are Hugo Pripp | | |

| Study trialist | Aleksi Reito |
|--------------------|----------------|
| Chief investigator | Antti Launonen |

#### **SECTION 2: INTRODUCTION**

# **Background**

In the ageing population, the proximal humerus fracture (PHF) is one of the most common fractures (2). In addition to the significant disability caused by PHF among older individuals, such fractures are also associated with a high economic impact (3). In general, the operative interventions and rehabilitation after a shoulder fracture are resource-consuming. The gender-specific fracture incidence for proximal humeral fractures for women in Sweden was 135 per 100000 person-years; in total, almost 10000 fractures were diagnosed in 2012 (4). The majority of PHFs are treated non-operatively and approximately 15%–33% of patients are treated surgically (5). Recent randomised controlled trials (RCTs) and metaanalyses have shown no difference in functional outcome between non-operative treatment and locking plate or hemi-arthroplasty (HA) in the treatment of PHF (6). However, operative treatment has a significantly higher risk of complications and reoperations of up to 30% (6). Originally, reverse total shoulder arthroplasty (RTSA) was used for osteoarthrosis in patients without cuff function to gain better functional outcomes. During the past decade, however, RTSA has gained popularity in the treatment of PHF. In a recent Medicare population analysis carried out between 2005 and 2012, the proportion of surgical procedures for PHF that were total shoulder arthroplasties (TSA) (of which RTSAs constituted 89% in 2011) increased from 3% to 17%, while the proportion of HA decreased from 42% to 24% during the same time period (5). There have been some systematic reviews based on case series and patient cohorts including one RCT that compared HA and RTSA. The results are equivocal; RTSA resulted in better functional outcomes compared with HA in some studies, with no difference seen in others (7, 8). In the RCT, the complication rate in the HA group was significantly higher than in the RTSA group (24% vs 10%, respectively). However, an arthroplasty registry analysis including 10844 operations (6658 TSA and 4186 RTSA) showed the RTSA postoperative complication rate to be 22% at 2 years (9). Currently, there are no RCTs comparing RTSA to non-operative treatment after PHF. The current literature discourages the operative treatment of PHF with locking plate or HA, and there is no evidence that favors surgery over non-operative treatment (6). In spite of the

substantial costs and lack of evidence supporting the effectiveness of RTSA for PHF, it has become the accepted standard of care in the USA. Therefore, there is an urgent need for high-quality RCTs that compare RTSA with non-operative treatment.

# Objectives and endpoint

### **SECTION 3: STUDY METHODS**

#### **Trial Design**

This was a prospective, superiority, single-blinded, randomised, controlled, multicentre and multinational trial that compared RTSA and non-operative treatment in proximal humerus fractures in patients aged 65–85 years with displaced three-part and four-part fractures (B and C types) according to the recent AO/OTA 2018 revision.

The Statistical Analysis Plan (SAP) is reported in accordance with the "Guidelines for the Content of Statistical Analysis Plan in Clinical Trials" (10).

The Deltacon trial is registered at <a href="www.clincaltrials.gov">www.clincaltrials.gov</a> with the number NCT03531463. The primary ethical approval for the trial has been given by the Regional Committee for Medical and Health Research Ethics, South-East Authority, Norway (2018/476 REK sør-øst D, <a href="https://rekportalen.no/#hjem/home">https://rekportalen.no/#hjem/home</a>). All sites gained institutional approval before the start of the trial. All patients included in the trial and those who declined but were asked to take part in the follow-up cohort were asked to give written informed consent.

#### Randomisation

Patients were randomised using a random number matrix in a block allocation fashion, in blocks of 10. The blocks were stratified by age (65–75 years and >75 years) since age has been shown to associate with the main outcome measure. The treatment allocations from the matrix were acquired from an online randomisation system (website http:// randomize. net), where the researcher logged in after written consent and received the correct intervention. The randomisation system asked for stratified items: The hospital (site), gender and patient

age. Thereafter, the allocation will be shown. The patient was randomised after written consent and before baseline assessments. The physician responsible for the intervention or treatment did not participate in any part of the collection of patient outcomes during the follow-ups.

# **Sample Size**

Assuming the effect size of a 14-point difference in the QuickDASH score and an SD (equal for both groups) of 26.8 points (from previous Olerud and MacDermid trials), the estimated sample size was 58 patients per group (delta=14, SD=26.8, alpha=0.05, power=0.8). With this age group, the estimate of loss in follow-up rate was set to 25% and resulted in a total of 154 patients in the trial. Total recruitment achieved 154 patients.

#### Framework

The overall objective of the trial was to determine whether surgical intervention results in a clinically and statistically significant better improvement compared to non-operative treatment on the short form of Disabilities of the Arm, Shoulder and Hand (Quick-DASH). The primary hypothesis is that surgical intervention produces better functional outcome and less pain compared to the non-operative treatment at 24 months.

#### **Estimands**

# Clinical question

Among patients aged 65–85 years with displaced 3- or 4-part proximal humerus fractures (AO/OTA 11-B and 11-C types) who meet the trial eligibility criteria, what is the effect of initial randomisation to RTSA versus non-operative treatment on shoulder-related disability at 24 months?

# Primary estimand components

| Component | Specification |
|---|---|
| Treatment | Initial randomised assignment to RTSA versus non-operative treatment (exercise), |
| condition | regardless of subsequent treatment changes (treatment policy for most intercurrent |
| | events, see Section 4.x.2). |
| Target | All randomized participants meeting the inclusion and exclusion criteria at |
| population | baseline (intention-to-treat population), aged 65-85 years with AO/OTA 11-B1.1, |
| | 11-B1.2, 11-C1.1, 11-C3.1 low-energy PHF types as defined in the protocol. |

| Variable | Short form Disabilities of the Arm, Shoulder and Hand (QuickDASH) score (0- |
|---|---|
| (endpoint) | 100, higher = greater disability) assessed at 24 months after randomisation. |
| Intercurrent | Death before 24 months, secondary surgery (including revision, conversion to |
| events | arthroplasty), crossover between treatment groups, additional non-protocol |
| | physiotherapy, and other changes in shoulder-related treatment after |
| | randomisation. |
| Strategy for | Treatment policy strategy for surgery/crossovers/other shoulder procedures; |
| intercurrent | treatment policy for additional non-protocol rehabilitation; composite strategy for |
| events | death (patients dying before 24 months assigned the worst possible QuickDASH |
| | score). |
| Population-level | Adjusted mean difference in QuickDASH score at 24 months between RTSA and |
| summary | non-operative treatment, estimated from the pre-specified linear mixed model, with |
| | 95% confidence interval. |
| Hypothesis | RTSA provides a clinically and statistically significant reduction (improvement) in |
| | QuickDASH score at 24 months compared to non-operative treatment. |

Analysis model corresponding to the primary estimand

The primary estimand will be estimated using the pre-specified linear mixed-effects model:

- Random effect: patient (to account for repeated measures).
- Fixed effects: treatment group, follow-up time (3 months, 12 months, 24 months), treatment-by-time interaction, study centre, baseline QuickDASH, and age.
- Primary contrast: adjusted mean difference in QuickDASH at 24 months between RTSA and non-operative treatment, obtained as estimated marginal means from the model.

This analysis yields an estimate of the primary estimand under the assumption that missing data are missing at random conditional on the included covariates (see Missing Data section).

# Secondary Estimands

For key secondary outcomes (VAS pain, grip strength, OSS, Constant Score, 15D, and reoperation/complication outcomes), estimands follow the same general structure:

- Treatment: randomised RTSA vs non-operative treatment (treatment policy).
- Population: all randomised eligible participants (ITT).
- Variables: respective secondary endpoints at prespecified time points (3, 12, 24 months).

- Intercurrent events: handled as per Section 4.x.3 (same as for primary).
- Summary measures:
  - For continuous outcomes: adjusted mean differences at 24 months from mixed models.
  - For binary outcomes: absolute risk differences at each time point from logistic regression with marginal effects.

A per-protocol estimand for the primary outcome will be defined as the effect of RTSA versus non-operative treatment among participants who adhered to their allocated initial treatment and had no major protocol deviations. This provides a sensitivity estimand complementary to the primary ITT estimand.

# Intercurrent Event Strategy

The table below specifies how each type of intercurrent event will be handled for the primary and key secondary estimands.

| Intercurrent event | Definition / examples | Implementation in analysis |
|---|---|---|
| Death before 24-month | Patient dies from any cause before | Patients who die before the 24-month |
| follow-up | the 24-month outcome can be | assessment will be considered as missing and |
| | obtained. | all data until death is included in the analyses. |
| Crossover from non- | Patient randomised to non- | Patient remains analysed in the originally |
| operative to RTSA or | operative treatment undergoes | allocated group (non-operative) for ITT. All |
| other surgery | RTSA or other shoulder surgery | available QuickDASH measurements, |
| | during follow-up. | including post-surgery, are used in the mixed |
| | | model. Crossover is documented and will be |
| | | explored in per-protocol (as-treated) sensitivity |
| | | analyses. |
| Failure to receive | Patient randomised to RTSA does | Patient remains in the RTSA group for ITT |
| allocated RTSA (no | not receive RTSA (e.g. surgery | analysis. All available outcomes are analysed |
| surgery or different | cancelled, different procedure | as randomised. A per-protocol analysis will |
| procedure) | performed, or major deviation | exclude or reclassify such patients according |
| | from planned implant). | to predefined PP criteria. |
| Revision surgery or | Any reoperation on the index | Outcomes collected after revision or secondary |
| secondary surgery after | shoulder (e.g. revision | surgery are included as observed, reflecting the |
| the index procedure or | arthroplasty, conversion to RTSA, | overall effect of the initial treatment strategy, |
| initial care | hardware removal, re-fixation). | including complications and subsequent |
| | | interventions. |

| Additional or intensified | Any non-protocol variation in | Considered part of real-world management |
|---|---|---|
| physiotherapy / | physiotherapy intensity, duration | following the initial treatment assignment; |
| rehabilitation | or setting after randomisation. | outcomes included as observed. No adjustment |
| | | will be made specifically for post- |
| | | randomisation physiotherapy use or adherence |
| | | in the primary analysis, but may be described |
| | | descriptively. |
| Permanent | Patient becomes institutionalised, | Where feasible, outcome data may be collected |
| institutionalisation or | develops severe comorbidity, or is | by mail or telephone. If no data are obtained at |
| severe decline preventing | otherwise unable to attend | 24 months, the mixed model will use available |
| clinic attendance | physical follow-up, but remains | earlier measurements under MAR assumption. |
| | alive. | |
| Withdrawal of consent | Patient withdraws consent to | Previously collected data will be included; no |
| for further data collection | attend further visits but allows use | further data collected. Mixed model estimates |
| (but permission to use | of already collected data. | will rely on available data assuming MAR. |
| prior data) | | |
| Withdrawal of consent | Patient withdraws consent and | All data from that participant will be excluded |
| including use of prior | requests deletion/non-use of prior | in accordance with applicable regulations and |
| data | trial data. | ethics. This change will be documented, and |
| | | the effective analysis population will be |
| | | reduced accordingly. |
| Discovery of ineligibility | Patient is found after | For ITT estimand, such patients remain |
| after randomisation | randomisation not to meet one or | included and analysed as randomised. For the |
| | more inclusion/exclusion criteria | per-protocol estimand, these participants will |
| | (e.g., misclassified fracture type). | typically be excluded (see detailed PP |
| | | definition). |

# Statistical interim analysis and stopping guidance

The external trial board had access to interim data and carried out the interim analysis after recruiting half of the patients. The report concentrated on the number of AEs and provided a recommendation on whether or not the trial should proceed. The board assessed the complication rates and compared them to the expected rates published in the available literature. An unexpectedly high rate of complications in either group would have indicated the end of the randomisation.

Date: 26.12.25

Version: 1.3.2

They advised the trial to continue. AEs and serious adverse events (SAEs) will be reported

according to the guidelines provided by the Consort Group.

AE is defined in 3 categories (mild, moderate, severe) as follows:

1. For the RTSA intervention group, the primary focus will be postoperative deep infections

requiring revision surgery, instability, periprosthetic fracture, radiographic early signs of

loosening (within 2 years of the surgery) of the humeral stem or notching of the scapula neck.

2. For the non-operative group, the primary focus will be on the rate of secondary surgery for

any reason (eg, non-union, symptomatic avascular head necrosis, osteoarthrosis).

Both groups were monitored for SAE during the first four weeks after discharge for

embolism (cardiac or brain) or death. The research nurse or physiotherapist filled out AE and

SAE forms at 3 months control, if needed. At the halfway point of the trial (50% of patients

recruited), an independent steering committee evaluated the complication rates and correlate

them to the expected rates published in the available literature.

Timing of final analysis

The final analysis for the primary outcome, the end scores on QuickDASH at 24 months, will

be performed after the last follow-up assessment at 24-months. The main publication of the

trial will be prepared when these data are available.

In addition, papers on 5- and 10-years follow-up will be performed, when these follow-up

assessments are available.

Timing of outcome assessments

The trial consists of six time points; baseline, 12-weeks, 12-months, 2 years, 5 years and 10

years. An overview of the assessments and procedures has been presented in the protocol.

**SECTION 4: STATISTICAL PRINCIPLES** 

Confidence intervals and P values

Date: 26.12.25

Version: 1.3.2

For the primary outcome the statistical tests will be two-sided and a p-value <0.05 will be

considered statistically significant. Confidence intervals will be 95% (95% CI) and two-

sided.

No adjustments for multiplicity were made. For the secondary outcomes, p-values will be

downplayed when interpreting the results. Secondary outcome are exploratory.

**Analysis populations** 

The primary analysis will be based on the Intention to Treat (ITT) principle. Patients

allocated to a treatment group (RTSA or exercise) should be followed up, assessed and

analysed as members of that group, regardless of their adherence to the planned course of

treatment. Per-protocol analysis population was defined as patients meeting protocol

requirements, receiving either RSTA or nonoperative treatment, regardless of primary

allocation, and not lost to follow-up immediately after randomisation (provided outcome data

at least 1 time-point).

**Changes from the Protocol** 

We have modified the primary statistical analysis from what was specified in the original

protocol. The protocol originally described univariable comparisons at each time point.

However, the updated analysis employs a linear mixed model, which more appropriately

accounts for repeated-measures data. Dichotomous outcomes will still be analysed at each

time point as originally planned, but the treatment effect will be estimated as the difference in

proportions derived from marginal estimates of a logistic model.

The primary analyses described in the original protocol are now considered supplemental

analyses.

The original protocol contained a typographical error in the sample size calculation (incorrect

loss to follow-up). The corrected calculation is presented in this SAP and corresponds to the

intended assumptions described in the protocol.

**SECTION 5: TRIAL POPULATION** 

Screening data

At all hospitals patients eligible for treatment were screened for the inclusion and exclusion criteria. If they fulfilled the criteria, they were invited to participate. The number of patients who did not meet the criteria and the reason for ineligibility will be reported in a CONSORT flow chart. There were no pre-randomization withdrawals.

# **Eligibility**

The following criteria was used throughout the study for patient selection.

- Inclusion criteria:
  - Low-energy AO/OTA group 11-B1.1, 11-B1.2 and 11-C1.1, 11-C3.1 (11). Both B and C type includes the subgroups: displaced,<sup>2</sup> impacted<sup>3</sup> or non-impacted<sup>4</sup> from the universal modifiers list.
- Exclusion criteria:
  - o Radiographic
    - Mal-inclination less than varus 30° or valgus 45°.
    - Less than 50% contact between head fragment and metaphysis/diaphysis.
    - Head split fractures (group 11-C3.2 and 11-C3.3) with >10% of the articular surface in the main head fragment.
    - Dislocation or fracture dislocation of the gleno-humeral joint.
    - Pathological fracture.
    - Glenoid abnormality (retroversion, >15°; glenoid fracture; cuff arthropathy).

#### o General

- Refuses to participate in the study.
- Aged <65 years or >85 years.
- Serious poly-trauma or additional surgery.
- Non-independent, drug/alcohol abuse or institutionalized (low cooperation).
- Contraindications for surgery (severe cardiovascular, pulmonal or neurological comorbidity).
- Does not understand written and spoken guidance in local languages.
- Previous fracture with symptomatic sequelae in either shoulder.
- Patients living outside the hospital's catchment area.

Recruitment

The CONSORT flowchart will present the number of patients screened, excluded (with

reasons), eligible for inclusion, randomized, receiving allocated treatment, withdrawals (with

reasons), lost to follow-up (with reasons), included in the ITT analysis, included in the per

protocol analysis.

Withdrawal/follow-up

Throughout the trial period, the included patients were allowed to withdraw from the study at

any time. Participants who decided to withdraw will be encouraged to continue in the study

as if they have received the intervention.

**Baseline patient characteristics** 

Baseline characteristics will be presented. Categorical variables will be presented as numbers

and percentages. Continuous variables will be presented as mean with standard deviation

(SD), if normally distributed and ad median with interquartile range (IQR) if not normally

distributed. No tests of significance will be conducted for the baseline characteristics,

imbalances of importance will be noted. Baseline and follow-up values for the primary and

secondary outcomes will be presented as part of the analysis.

From the baseline variable, age and baseline QuickDASH were included for adjustment in the

analyses. Missing baseline data is reported.

**SECTION 6: ANALYSIS** 

**Outcome definitions** 

**QuickDASH** 

The primary outcome will be presented as the 24-month adjusted mean difference.

QuickDASH is a valid and reliable patient-reported questionnaire assessing shoulder pain and

function with 11 items. The final score is between 0 to 100, where higher score indicates

greater disability.

Secondary outcomes

General visual analogue scale (VAS) for pain, grip strength, the Oxford Shoulder Score (OSS), the Constant score (CS) and the number of reoperations and complications. Quality of life will be assessed with 15-D. Difference in treatment costs between the groups will be calculated and health economic analysis performed.

# **Analysis methods**

The primary analysis method for QuickDASH will be a linear mixed model. The patient is included as a random factor. Study group and follow-up assessments (3 months, 1 year, 2 years) will be included as a fixed factor. Study centre, baseline QuickDASH and patient age will also be included as fixed factors. The main model will include the interaction between the study group and the follow-up assessment. Primary treatment effect at 2 years will be estimated as the estimated marginal means between the study group from time-spesific contrast. Similar estimates will be obtained for 3 months and 1 year also. Similar analysis will be done for key secondary outcomes VAS pain, VAS grip strength, OSS, CS and 15D. Results will be presented with 95% CIs.

For categorical variables we will estimate the group absolute risk difference using a logistic regression based on marginal effects. Separate models will be run at each follow-up timepoints. Logistic models include study group and patient age as adjusting covariates.

No residual diagnostics were done as LMM is robust against normality violations (12). Baseline imbalances were addressed including age and baseline QuickDASH in the LMM analysis. Age is the single most important variable affecting the outcome.

#### Missing data

As stated above, imputations will not be applied in this study due to the repeated mixed model analysis. We assume missing at random (MAR) model. Each randomized patient will be included in the intention-to-treat analysis with the collected data. In an attempt to collect data from all randomized patients, participants deciding to withdraw from the study, are still encouraged to attend the follow-up test.

# Additional analyses

For primary and key secondary outcomes an additional analysis will be done with a crude between-group comparison. For continuous variables we will assess the study group difference using Welch t-test at each time point as a supplementary analysis. Categorical variables will be compared using Fisher exact test for 2x2 tables and Chi-squares test for other comparisons.

The subgroup analyses for the primary outcome will be done according to following variables: of age (per stratification), sex, fracture group, smoking and ASA class. These analyses are as stratified not using interaction analysis. No adjustment for multiplicity is done and all analyses are purely exploratory.

Additional analyses will be performed with the purpose of testing the robustness of the intention-to-treat analysis, including a per-protocol analysis for the primary outcome; Crossover patients are defined as patients allocated to the non-operative group who undergo RSA during follow-up or patients allocated to surgery, but who do not undergo the procedure to any reason. Between operated patients, a sensitivity analysis will be conducted comparing different models of prostheses.

#### Harms

Adverse and serious adverse events will be presented as numbers and percentages for each event.

### Statistical software

All statistical analysis will be made using the latest R software and/or Stata

- 1. Launonen AP, Fjalestad T, Laitinen MK, Lahdeoja T, Ekholm C, Wagle T, et al. Nordic Innovative Trials to Evaluate osteoPorotic Fractures (NITEP) Collaboration: The Nordic DeltaCon Trial protocol-non-operative treatment versus reversed total shoulder arthroplasty in patients 65 years of age and older with a displaced proximal humerus fracture: a prospective, randomised controlled trial. BMJ Open. 2019;9(1):e024916.
- 2. Launonen AP, Lepola V, Saranko A, Flinkkila T, Laitinen M, Mattila VM. Epidemiology of proximal humerus fractures. Archives of osteoporosis. 2015;10(1):209.
- 3. Fjalestad T, Hole MO, Jorgensen JJ, Stromsoe K, Kristiansen IS. Health and cost consequences of surgical versus conservative treatment for a comminuted proximal humeral fracture in elderly patients. Injury. 2010;41(6):599-605.

4. Sumrein BO, Huttunen TT, Launonen AP, Berg HE, Fellander-Tsai L, Mattila VM. Proximal humeral fractures in Sweden-a registry-based study. Osteoporos Int. 2016.

- 5. Han RJ, Sing DC, Feeley BT, Ma CB, Zhang AL. Proximal humerus fragility fractures: recent trends in nonoperative and operative treatment in the Medicare population. J Shoulder Elbow Surg. 2016;25(2):256-61.
- 6. Handoll HH, Elliott J, Thillemann TM, Aluko P, Brorson S. Interventions for treating proximal humeral fractures in adults. Cochrane Database Syst Rev. 2022;6:CD000434.
- 7. Bonnevialle N, Tournier C, Clavert P, Ohl X, Sirveaux F, Saragaglia D, et al. Hemiarthroplasty versus reverse shoulder arthroplasty in 4-part displaced fractures of the proximal humerus: Multicenter retrospective study. Orthop Traumatol Surg Res. 2016;102(5):569-73.
- 8. Khan WS, Longo UG, Ahrens PM, Denaro V, Maffulli N. A systematic review of the reverse shoulder replacement in rotator cuff arthropathy, rotator cuff tears, and rheumatoid arthritis. Sports Med Arthrosc. 2011;19(4):366-79.
- 9. Villacis D, Sivasundaram L, Pannell WC, Heckmann N, Omid R, Hatch GF, 3rd. Complication rate and implant survival for reverse shoulder arthroplasty versus total shoulder arthroplasty: results during the initial 2 years. J Shoulder Elbow Surg. 2016;25(6):927-35.
- 10. Gamble C, Krishan A, Stocken D, Lewis S, Juszczak E, Dore C, et al. Guidelines for the Content of Statistical Analysis Plans in Clinical Trials. Jama. 2017;318(23):2337-43.
- 11. Kellam JF, Meinberg EG, Agel J, Karam MD, Roberts CS. Introduction: Fracture and Dislocation Classification Compendium-2018: International Comprehensive Classification of Fractures and Dislocations Committee. J Orthop Trauma. 2018;32 Suppl 1:S1-S10.
- 12. Arnau J, Bendayan R, Blanca MJ, Bono R. The effect of skewness and kurtosis on the robustness of linear mixed models. Behav Res Methods. 2013;45(3):873-9.